CLINICAL TRIAL: NCT06038903
Title: Evaluation of The Psychometric Properties of The Turkish Version of The Brief-Caffeine Expectancy Questionnaire (B-CaffeQ): An Adaptation Study in Recreationally Active Individuals
Brief Title: The Turkish Version Of The Brief-Caffeine Expectancy Questionnaire
Status: Completed | Type: Observational
Sponsor: Eskisehir Technical University (Other)
Responsible Party: Principal Investigator, Celil Kaçoğlu, Associated profesor, Eskisehir Technical University
Other Study IDs: EskisehirTU-SBF-CK-02
Record Dates: First submitted 2023-09-08; First posted 2023-09-15 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Caffeine; Adaptation; Expectations; Language
Keywords: expectation; caffeine; Brief-Caffeine Expectancy Questionnaire; Language adaptation study
MeSH Terms: conditions — Language

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- EFA group: This group for exploratory factor analysis (EFA)
  Interventions: Other: caffeine consumption expectation
- CFA group: This group for confirmatory factor analysis (CFA)
  Interventions: Other: caffeine consumption expectation

INTERVENTIONS:
Other: caffeine consumption expectation — The group to which the Short-form caffeine expectation questionnaire (B-CaffeQ) was applied, which evaluated the expectations from caffeine consumption.

SUMMARY:
Caffeine is a psycho-active substance that is widely consumed in the world. It is seen that its widespread consumption is related to expectancies of consumption as well as cultural factors. Recreationally active individuals may have various expectations from caffeine consumption in line with their lifestyles and goals such as physical, social and/or other aspects. It can be stated that caffeine consumption expectancies have an important role in the process of evaluating consumption patterns. However, in the literature it seems to be very limited information about expectancies related to caffeine consumption. In this direction, the aim of the research was to test the compatibility of Brief-Caffeine Expectancy Questionnaire (B-CaffeQ) to Turkish culture and language. In the study, data will be collected from two separate participant groups and going to analysis. To reveal the structure on the first group (n=250-300 approx.) data, Exploratory Factor Analysis (EFA), and to verify the structure on the second group (n=313) data, Confirmatory Factor Analysis (CFA) will be used. Reliability will be assessed by performing test-retest and internal consistency analyzes on both the two data groups.

DETAILED DESCRIPTION:
INTRODUCTION

Caffeine (1,3,7-trimethylxanthine) is most commonly found in coffee as the main pharmacologically active ingredient. In general, brewed coffee has the highest content among foodstuffs containing caffeine. Coffee (230-250ml), depending on the preparation method, the type of beans, roasting, grinding type and brand, contains 35-250 mg of caffeine while tea (150 ml) 24-50 mg, cola drinks (180 ml) 15-30 mg, cocoa (150 ml) 2-7 mg, chocolate (28 g) 1-36 mg, and the foods containing chocolate mostly contain less than 15 mg caffeine.

Doses of up to 300-400mg per day in healthy adults (19 and over) are specified as safe upper limit without any harmful effects. This amount corresponds to 4-5 cups of medium coffee. However, it is stated that caffeine consumption equal to 6 cups of dark coffee generally does not cause any side effects. It is stated that the daily limit for adolescents and children is 100 mg and this limit should not be exceeded. However, coffee is not the only source of caffeine, and other sources caffeine consumed should also be taken into account.

The average daily caffeine consumption in Turkey for adolescents and children aged 15 and below is an average of 197 mg and 202 mg for 18 and older. The source of caffeine for adolescents is mostly tea, carbonated soft drinks and instant coffee consumption. Average daily caffeine consumption in adult working individuals is 247 mg, and this is due to the consumption of carbonated soft drinks, chocolate, instant coffee, respectively. It is seen that 20% of university students who consume caffeine have an average daily consumption of 250 mg and above, and this mostly due to the consumption of tea, coffee, Turkish coffee, carbonated soft drinks and chocolate. In USA, while the main source of caffeine is coffee for the age of 18 and above, it is caffeine-containing soft drinks for the age of 2-17.

There is evidence that some individuals' expectancies of caffeine's effects on physical performance and mood may affect the magnitude of these effects. There are studies showing that caffeine anticipation effect affects mood, attention, and vitality. In the case of caffeine expectancy, placebo administration stimulates changes in the dopaminergic system in the brain. The neurobiological mechanisms of caffeine and placebo caffeine were similar in the brain, but somewhat more limited in placebo caffeine. It is stated that the expectancy of the individual may manage the placebo effect and accordingly, the expected effect of caffeine or the drug consumed may change the response to placebo. Beyond the pharmacological effects of a drug, an individual's expectancies of it may also contribute to the intensive experiences of the drug in question. The fact that individuals who are told they had decaffeinated coffee but are given caffeine perform worse than those who do not consume caffeine, support the view that the pharmacological effects of caffeine act synergistically with anticipation. In addition, it has been stated that the effects caused by caffeine withdrawal may also be caused by the negative expectancies (nosebo) of an individual. These results provided evidence that the subjective and behavioral effects of caffeine consumption may be positive or negative depending on the individual's expectancies from caffeine. These expectancies may arise from the individual's previous experiences with caffeine. The effects of caffeine depend on the individual's expectancies, so if the individual consumes a beverage expecting that it has caffeine in it, these expectancies may be generalized as placebo conditions. In placebo studies, it is stated that one of the factors that cause an individual to respond to a treatment may be caused by the type of individual who may respond to treatment via expectancies. In other words, this view is not specific to the treatment of the practice applied, rather that the response may be shaped according to the expectancies of the individual, that expectancies may cause a placebo (or nosebo) effect. When there is confidence in the drug effect of a drug in a particular activity, an expectancy of a specific behavioral effect of that drug may also be formed. Based on expectancies about the effects of caffeine, the behavioral response to this drug derivative can be predicted. However, this expectancy theory is insufficient to explain the fact that some individuals without expectancies not showing stimulating effects when they consume caffeine for the first time. There are other studies which do not observe expectancy affects in caffeine consumption, suggesting placebo and expectancy effects are caused by introspection. The results showed that both pharmacological and expectancy factors affect the actual and expectancy effects of caffeine in an individual's behaviour.

Some of the performance enhancing effects of caffeine appear to be linked to expectancies. Since the bitter taste of caffeine may act as a signal that caffeine has been consumed, it seems possible that some anticipatory effects of caffeine consumption may be driven by this bitter taste. It is said that consuming 300-400 mg caffeine a day, equivalent of 3-4 cups of coffee daily, may have positive effects on the well-being of an individual and may partially improve mental-physical disorders. Performance increases were also observed with individuals who consume coffee regularly when they are given decaffeinated coffee. This suggests a caffeine related stimulus causes a caffeine related effect. This result also indicates, other features of coffee such as its smell and taste rather than caffeine itself, may also be effective in the development of these expectancies. It has been observed when these individuals who consume coffee regularly do not wish to consume caffeine yet want to benefit from its performance enhancement effects, decaffeinated coffee also creates a good effect on performance enhancement. In addition, the expectancy for the positive effects of caffeine consumption is an indicator of how much and how often caffeine will be consumed.

PURPOSE OF RESEARCH Since caffeine consumption is rather widespread in Turkey, it can be seen that an instrument to be used in research on caffeine consumption expectancies such as caffeine expectancy survey is needed. Accordingly, the purpose of this research is to adapt and verify the Breif-Caffeine Expectancy Questionnaire (B-CaffeQ) which has been developed by Kearns et al. (2018) and consists of seven dimensions: withdrawal / dependence, energy / work enhancement, appetite suppression, social / mood enhancement, physical performance enhancement, anxiety / negative physical effects, and sleep disturbance, to Turkish culture and language.

METHODOLOGY Research model

This research model includes a methodological process in which the Brief-Caffeine Expectancy Questionnaire is evaluated through the validity and reliability analysis of the Turkish language and culture. This process includes some steps will be deemed necessary for the adaptation of the questionnaire. These stages will be followed in the following order:

* Survey translation.
* Evaluating the items and making the necessary corrections.
* Testing the items.
* Creating the initial form of the questionnaire.
* Implementation of the survey.
* Conducting analyses.
* Finalizing the questionnaire.
* Examination of the measurement model.
* Reporting of the process.

Research group The participants in this study are recreationally active individuals. Data will be collected from two different groups for validity and reliability assessments. Data will be obtained from the first group, in which the processes related to Exploratory Factor Analysis (EFA) will be carried out, and the processes related to Confirmatory Factor Analysis (CFA) will carry out with the data collected from the second group. Groups consist of participants will select by the purposive sampling. For the purpose of this research, individuals who consume products containing caffeine such as coffee, tea, and soft drinks constitute the research group. Accordingly, data will collect from 250-300 (aprroximately) participants for EFA process and from 30 participants for CFA process.

Ethical clearance The study protocol was approved by the Scientific Research and Publishing Ethics Committee of Eskisehir Technical University (Decree number: E-87914409-050.03.04-8971).

Data collection tool and technique During the data collection phase, a questionnaire form consisting of three parts will use. In the first part, explanations about the research and caffeine containing product information which the participant based their answers on included. In the second part of the questionnaire, Brief-Caffeine Expectancy Questionnaire, which is a simplified version of the caffeine expectancy questionnaire developed by Huntley and Juliano, will be included. This questionnaire, whish has been simplified by Kearns et al. (2018) by carrying out validity and reliability studies, has a 7-factor structure, consisting of 20 articles. The rating of this questionnaire, which was created in six Likert type, was defined as "1 = Strongly Disagree" to "6= Strongly Agree". In the last part of the questionnaire, there will be questions from which the demographic information of the participants such as age, gender, educational status, etc. obtain.

Aforementioned questionnaire form will be prepared on an online platform and the connection link will be provided. This link will be conveyed to participants through posts shared on these social media accounts.

Language equivalence In the process of adapting B-CaffeQ to Turkish language and culture, back translation method will be used in order to provide language equivalence. Accordingly, both the English to Turkish and Turkish to English translations will made independently by two different linguists who are adept in both languages and cultures. Finally, the articles will translate back into English and compare with their original forms.

Data analysis EFA will use in order to determine what kind of a structure pattern the survey constitutes in Turkish language and culture. CFA will use to test the accuracy of the structure resulting from EFA. Reliability tests of the questionnaire will perform through Cronbach Alpha coefficient and test-retest analysis.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 60
* Physical health individuals

Exclusion Criteria:

* Heart disease
* Using of pacemaker
* Epilepsy
* Transient ischemic attack
* Stroke or similar nervous disorders
* Psychiatric disease
* Cardio-pulmonary diseases
* Pregnancy
* Drug using that affect the heart rate and blood pressure
* Systemic, neuroplastic, inflammation disorders

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Physically active, physiologically healthy and routinely caffeine consumer male and females between 18-60 ages.
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2023-09-08 (Actual); Primary Completion 2023-10-10 (Actual); Study Completion 2023-10-15 (Actual)

PRIMARY OUTCOMES:
the Breif-Caffeine Expectancy Questionnaire (B-CaffeQ) | two weeks
  Brief-Caffeine Expectancy Questionnaire, which is a simplified version of the caffeine expectancy questionnaire developed by Huntley and Juliano (2012), will be included. This questionnaire, whish has been simplified by Kearns et al. (2018) by carrying out validity and reliability studies, has a 7-factor structure, consisting of 20 articles (Huntley & Juliano, 2012; Kearns et al., 2018). The rating of this questionnaire, which was created in six Likert type, was defined as "1 = Strongly Disagree" to "6= Strongly Agree". In the last part of the questionnaire, there will be questions from which the demographic information of the participants such as age, gender, educational status, etc. obtaine.

CONTACTS AND LOCATIONS:
Overall Officials: celil kaçoğlu, assoc. prof., Principal Investigator — Eskişehir Tecnical University
Locations (1):
- Eskişehir Technical University, Eskişehir, Tepebaşı, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No